CLINICAL TRIAL: NCT04939272
Title: A Phase 1/2 Study of Copanlisib and Venetoclax in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Copanlisib and Venetoclax for the Treatment of Relapsed or Refractory Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22043; NCI-2021-03219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22043 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-06-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — copanlisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (copanlisib hydrochloride, venetoclax) (Experimental): Patients receive copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15, and venetoclax PO QD on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Copanlisib will be given at 30mg, 45mg, or 60 mg depending on the assigned dose level. Venetoclax will have a weekly dose ramp up from 20mg, 50mg, 100mg, 200mg, and then 400mg thereafter.
  Interventions: Drug: Copanlisib Hydrochloride; Drug: Venetoclax

INTERVENTIONS:
Drug: Copanlisib Hydrochloride — Patients receive copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 for each cycle.
  Copanlisib will be given at 30mg, 45mg, or 60 mg depending on the assigned dose level.
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
Drug: Venetoclax — Patients receive venetoclax PO QD on days 1-28 for each cycle. Venetoclax will have a weekly dose ramp up in cycle one from 20mg, 50mg, 100mg, 200mg, and then 400mg daily thereafter starting from cycle 2.
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial studies the side effects, best dose, and effectiveness of copanlisib and venetoclax in treating patients with mantle cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Copanlisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving copanlisib and venetoclax may help treat patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety, tolerability, and the maximum tolerated dose (MTD) of copanlisib hydrochloride (copanlisib) and venetoclax in patients with relapsed/refractory (R/R) mantle cell lymphoma (MCL). (Phase 1) II. To estimate the efficacy (as measured by overall rate of response [ORR]) of copanlisib in combination with venetoclax in patients with R/R MCL. (Phase 2)

SECONDARY OBJECTIVES:

I. To characterize the safety profile of copanlisib in combination with venetoclax in patients with R/R MCL. (Phase 2) II. To evaluate duration of response (DOR) and progression-free survival (PFS) associated with combined administration of copanlisib/venetoclax. (Phase 2) III. To evaluate an overall survival (OS) associated with combined administration of copanlisib/venetoclax. (Phase 2) IV. To characterize the pharmacokinetics (PK) profile of copanlisib and venetoclax. (Phase 2)

EXPLORATORY OBJECTIVES:

I. Evaluate the emergence of resistant clones, as determined by the presence of novel mutations and expression of BCL2 family proteins.

II. Characterize the T-cell population balance in patients treated with copanlisib/venetoclax.

OUTLINE: This is a phase I, dose-escalation study of copanlisib hydrochloride, followed by a phase II study.

Patients receive copanlisib hydrochloride intravenously (IV) over 1 hour on days 1, 8, and 15, and venetoclax orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Life expectancy >= 3 months (per physician assessment)
* Ability to take oral medication
* Pathologically confirmed MCL, with documentation of monoclonal B cells showing one of the following:

  * Overexpression of cyclin D1 in association with other relevant markers (e.g., CD19, CD20, PAX5, CD5), OR
  * Chromosomal translocation t(11;14)(q13; q32), as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR)
* Documented failure to achieve at least partial response (PR) with, or documented disease progression after the most recent treatment regimen
* At least 1 prior treatment regimen for MCL which either included chemo-immunotherapy or a targeted agent (i.e., ibrutinib) administered for at least 2 cycles
* Have radiologically measurable lymphadenopathy or extranodal lesion, (defined as >= 1 lesion that measures >= 2.0 cm in the longest diameter), or splenomegaly, or bone marrow involvement with or without malignant lymphocytosis
* Absolute neutrophil count (ANC) >= 1,000/mm^3 without bone marrow involvement or ANC >= 500/mm^3 with bone marrow involvement (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 50,000/mm^3 without bone marrow involvement or platelets >= 30,000/mm^3 with bone marrow involvement (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment
* Total bilirubin =< 2 x upper limit of normal (ULN) (unless has Gilbert's disease or documented liver/biliary involvement by the lymphoma) (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Left ventricular ejection fraction (LVEF) >= 45% (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Lipase =< 1.5 ULN (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Glycosylated hemoglobin (HbA1c) =< 8.5% (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (to be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 30 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only) without an alternative medical cause.

Exclusion Criteria:

* Concurrent enrollment in another therapeutic investigational study
* Prior treatment with venetoclax (or other investigational small molecule BCL2 inhibitors) or with copanlisib
* Prior allogeneic stem cell transplant
* Prior therapeutic intervention with any of the following:

  * Therapeutic anticancer antibodies within 2 weeks
  * Radio- or toxin-immunoconjugates within 10 weeks
  * All other chemotherapy, radiation therapy within 30 days prior to initiation of therapy
  * Targeted therapy within 6 half-lives
* Vaccinated with live vaccines within 4 weeks of the first dose of study drug
* Systemic continuous corticosteroid therapy at a daily dose higher than 20 mg prednisone or equivalent is not allowed. Participants may be using topical or inhaled corticosteroids
* Concurrent administration of medications or food that are strong inhibitors or inducers of CYP3A4 taken within 7 days of starting study treatment
* Current evidence of central nervous system involvement by the lymphoma
* Uncontrolled active systemic infection
* Unresolved toxicities (except alopecia) from prior anticancer therapy (including radiation) that have not resolved to grade =< 1 (per Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0), or to the levels dictated in this protocol
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection

  * Participants who are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., breast, cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy or hormonal therapy
* Major surgery within 4 weeks of the first dose of study drug
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months of screening
* Uncontrolled arterial hypertension despite optimal medical management
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function, such as patients requiring oxygen supplementation
* Uncontrolled diabetes mellitus despite optimal medical management (per investigator's opinion)
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 3 months before the start of study medication
* Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (Phase I) | Up to end of cycle 2 (1 cycle = 28 days)
  Toxicities will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall response rate (Phase II) | Up to 2 years
  Defined as the proportion of response-evaluable participants that achieve a best response of either complete response (CR) or partial response (PR) during protocol therapy. Will be estimated along with the 2-sided 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Duration of response | Time from the first achievement of PR or CR to time of progressive disease, start of non-protocol anti-lymphoma therapy, or death, whichever earlier, assessed up to 2 years
  Will be estimated using the Kaplan-Meier product-limit method along with the Greenwood estimator of standard error; 95% confidence interval for the survival timepoint estimates will be constructed based on the log-log transformation. Median survival time will be estimated when available.
Progression-free survival | From start of protocol treatment to time of disease relapse/progression, or death due to any cause, whichever occurs earlier, assessed up to 2 years
  Will be estimated using the Kaplan-Meier product-limit method along with the Greenwood estimator of standard error; 95% confidence interval for the survival timepoint estimates will be constructed based on the log-log transformation. Median survival time will be estimated when available.
Overall survival | From start of protocol treatment to time of death due to any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier product-limit method along with the Greenwood estimator of standard error; 95% confidence interval for the survival timepoint estimates will be constructed based on the log-log transformation. Median survival time will be estimated when available.
Incidence of adverse events | Up to 90 days after completion of treatment
  Toxicity and adverse events will be recorded using the NCI CTCAE 5.0 scale. Safety and tolerability of copanlisib in conjunction with venetoclax will be summarized for all patients (evaluable for toxicity) combined and by dose level (if patients were treated at both dose level [DL]1 and DL-1). Adverse events will be tabulated and summarized by major organ category, grade, and drug attribution. Severe adverse event specific incidence and exact 95% confidence interval will be provided where necessary/appropriate.
Plasma pharmacokinetics (PK) of copanlisib (Cmax) | From 30 minute before Copanlisib on cycle 2 day 15 through 24 hours after (Each cycle is 28 days)
  Maximum plasma concentration (Cmax).
Plasma pharmacokinetics (PK) of copanlisib (AUC) | From 30 minute before Copanlisib on cycle 2 day 15 through 24 hours after.(Each cycle is 28 days)
  Area under the Curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Danilov, Principal Investigator — City of Hope Medical Cneter
Locations (1):
- City of Hope Medical Center, Duarte, California, United States